CLINICAL TRIAL: NCT06071104
Title: Next Generation Cataract Surgery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTV678-E002
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cataract
Keywords: Anterior segment ophthalmic surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- UNITY VCS (Experimental): Anterior segment ophthalmic surgery performed with UNITY VCS
  Interventions: Procedure: Anterior segment ophthalmic surgery; Device: UNITY VCS

INTERVENTIONS:
Procedure: Anterior segment ophthalmic surgery — Cataract surgery during which the crystalline lens (often cloudy) is broken into small pieces and gently removed from the eye with suction (phacoemulsification)
Device: UNITY VCS — UNITY Vitreoretinal Cataract System (VCS) with console, remote control, foot controller, UNITY Cataract FMS Pack, and UNITY Anterior Vitrectomy Kit

SUMMARY:
The purpose of this study is to obtain device-specific safety and performance clinical data to support marketability in Europe and to collect user preference data.

DETAILED DESCRIPTION:
Subjects will attend a screening visit (Day -60 to Day 0), a surgery visit (Day 0), and 3 post-surgical visits (Day 1, Week 1, Month 1) for an overall individual duration of up to 3 months. One eye (study eye) will be treated. This study will be conducted in the United States.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an IRB/IEC approved Informed Consent form.
* Willing and able to attend all scheduled visits as required by the protocol.
* Clinically documented diagnosis of age-related noncomplicated cataract.
* Eligible to undergo primary hydrophobic acrylic intraocular lens implantation into the capsular bag.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Women of childbearing potential as defined in the protocol.
* Planned postoperative procedures during the course of the study in the operative eye.
* Previous intraocular or corneal surgery in the operative eye.
* Diagnosis of glaucoma or ocular hypertension (IOP > 21 mmHg) in the operative eye.
* Other protocol-defined exclusion criteria may apply.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD Surgical, Study Chair — Alcon Research, LLC
Locations (4):
- United States (4):
  - Gordon Schanzlin New Vision Institute, A TLC Laser Eye Center, San Diego, California
  - Miramar Eye Specialists Medical Group, Ventura, California
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Vance Thompson Vision, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 investigative sites located in the United States.
Pre-assignment Details: Of the 121 participants enrolled in the study, 13 were exited prior to attempted treatment. This reporting group includes all participants with attempted treatment (108).
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | UNITY VCS
Started (Attempted implantation) | 108; 108 eyes
Completed | 107; 107 eyes
Not Completed | 1; 1 eyes
Not completed — Non-ocular and non-device related adverse event | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All eyes with attempted use of the UNITY VCS (successful or aborted after contact with the eye)
Arm/Group | UNITY VCS
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (6.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 104
  Black or African American | 1
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 108

OUTCOME MEASURES:

1. Primary Outcome: Percent of 'Yes' Responses to the Binary Question: "Did UNITY VCS Anterior Segment Surgical Functionality Perform Per the Intended Use as Defined in Protocol Section 5.1?"
Description: As recorded by the surgeon on a user questionnaire based on Day 0 surgery experience. From Protocol Section 5.1, the intended use for UNITY VCS is to facilitate management of fluid as well as removal, cutting, and coagulation of ocular materials. One eye (study eye) contributed data to the analysis. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Day 0
Population: All Implanted Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of responses
Units Other Than Participants: eyes
Arm/Group | UNITY VCS
Number analyzed (Participants) | 107
Number analyzed (eyes) | 107
percentage of responses | 99.1 [94.9 to 100.0]

2. Secondary Outcome: Time From Incision Entry to Incision Closure
Description: The time from incision entry to incision closure was measured using a stopwatch and recorded in seconds. One eye (study eye) contributed data to the analysis. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Day 0 surgery
Population: All Implanted Analysis Set
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | UNITY VCS
Number analyzed (Participants) | 107
Number analyzed (eyes) | 107
seconds | 376.8 (117.22)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, up to approximately 3 months.
Description: AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the investigator. This analysis population includes all subjects/eyes with attempted use of the UNITY VCS (successful or aborted after contact with the eye). The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more reporting groups.
Groups:
- Pretreatment: AEs in this group occurred prior to treatment with UNITY VCS
- UNITYVCSstudyeye: AEs in this group occurred after attempted treatment with with UNITY VCS and include ocular events in the study eye. "At Risk" population is reported in units of eyes.
- UNITYVCSSystemic: AEs in this group occurred after attempted treatment with UNITY VCS and include overall systemic events as well as ocular events in the non-study eye. "At Risk" population is reported in units of subjects.
Arm/Group | Pretreatment | UNITYVCSstudyeye | UNITYVCSSystemic
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/108 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/108 | 2/108 | 3/108
Other Adverse Events (participants affected / at risk) | 0/108 | 0/108 | 0/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=108) | UNITYVCSstudyeye (N=108) | UNITYVCSSystemic (N=108)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lens extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT06071104/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT06071104/SAP_001.pdf